| _ | | | |
|-----|----------------|-----|-----|
| C+. | | T:+ | ı |
| 711 | ıdy | 111 | 10. |
| ~ | <i>a</i> • • • | | |

Effects of preoperative combined use of acetaminophen and ibuprofen on the control of pain following orthodontic treatment

Approved on: 4/19/2017 Last updated: 4/19/2017

NCT #03523988



## **INSTRUCTIONS**

- <u>If you are requesting a determination</u> about whether your activity is human subjects research or qualifies for exempt status, you may skip all questions except those marked with a . For example **1.1** must be answered.
- Answer all questions. If a question is not applicable to your research or if you believe you have already answered a question elsewhere in the application, state "NA" (and if applicable, refer to the question where you provided the information). If you do not answer a question, the IRB does not know whether the question was overlooked or whether it is not applicable. This may result in unnecessary "back and forth" for clarification. Use non-technical language as much as possible.
- To check a box, place an "X" in the box. To fill in a text box, make sure your cursor is within the gray text box bar before typing or pasting text.
- The word "you" refers to the researcher and all members of the research team, unless otherwise specified.
- For collaborative research, describe only the information that is relevant to you unless you are requesting that the UW IRB provide the review and oversight for your collaborators as well.
- You may reference other documents (such as a grant application) if they provide the requested information in non-technical language. Be sure to provide the document name, page(s), and specific sections, and upload it to **Zipline**. Also, describe any changes that may have occurred since the document was written (for example, changes that you've made during or after the grant review process). In some cases, you may need to provide additional details in the answer space as well as referencing a document.

| INDEX | | |
|---|---|---|
| 1 Overview | 6 Children (Minors) and Parental Permission | 10 Risk / Benefit Assessment |
| 2 Participants | 7 Assent of Children (Minors) | 11 Economic Burden to Participants |
| 3 International Research Setting | 8 Consent of Adults | 12 Resources |
| 4 Recruiting and Screening Participants | 9 Privacy and Confidentiality | 13 Other Approvals, Permissions, and Regulatory Issues |
| 5 <u>Procedures</u> | | |

### **1 OVERVIEW**

**Study Title:** 

Effects of preoperative combined use of acetaminophen and ibuprofen on the control of pain following orthodontic treatment

**1.1 Home institution**. Identify the home institution of the lead researcher as listed on the IRB application. Provide any helpful explanatory information.

In general, the home institution is the institution (1) that provides the researcher's paycheck and that considers him/her to be a paid employee, or (2) at which the researcher is a matriculated student. Scholars, faculty, fellows, and students who are visiting the UW and who are the lead researcher: identify your home institution and describe the purpose and duration of your UW visit, as well as the UW department/center with which you are affiliated while at the UW.

Note that many UW clinical faculty members are paid employees of non-UW institutions.

The UW IRB provides IRB review and oversight for only those researchers who meet the criteria described in the **POLICY: Use** of the UW IRB.

University of Washington - School of Dentistry

(1.2)Consultation history. Have you consulted with anyone at HSD about this study?

It is not necessary to obtain advance consultation. If you have: answering this question will help ensure that the IRB is aware of and considers the advice and guidance you were provided.



→ If yes, briefly describe the consultation: approximate date, with whom, and method (e.g., by email, phone call, in-person meeting).

**1.3** Similar and/or related studies. Are there any related IRB applications that provide context for the proposed activities?

Examples of studies for which there is likely to be a related IRB application: Using samples or data collected by another study; recruiting subjects from a registry established by a colleague's research activity; conducting Phase 2 of a multi-part project, or conducting a continuation of another study; serving as the data coordinating center for a multi-site study that includes a UW site.

Providing this information (if relevant) may significantly improve the efficiency and consistency of the IRB's review.



→ If yes, briefly describe the other studies or applications and how they relate to the proposed activities. If the other applications were reviewed by the UW IRB, please also provide: the UW IRB number, the study title, and the lead researcher's name.

**1.4** Externally-imposed urgency or time deadlines. Are there any externally-imposed deadlines or urgency that affect your proposed activity?

HSD recognizes that everyone would like their IRB applications to be reviewed as quickly as possible. To ensure fairness, it is HSD policy to review applications in the order in which they are received. However, HSD will assign a higher priority to research with externally-imposed urgency that is beyond the control of the researcher. Researchers are encouraged to communicate as soon as possible with their HSD staff contact person when there is an urgent situation (in other words, before submitting the IRB application). Examples: a researcher plans to test an experimental vaccine that has just been developed for a newly emerging epidemic; a researcher has an unexpected opportunity to collect data from students when the end of the school year is only four weeks away.

HSD may ask for documentation of the externally-imposed urgency. A higher priority should not be requested to compensate for a researcher's failure to prepare an IRB application in a timely manner. Note that IRB review requires a certain minimum amount of time; without sufficient time, the IRB may not be able to review and approve an application by a deadline.

No X Yes

→ If yes, briefly describe the urgency or deadline as well as the reason for it.

The proposed activity is to be completed as part of a 4<sup>th</sup> year dental student research-focused curriculum. The dates for the student to conduct the clinical trials range from March 27<sup>th</sup> to June 16<sup>th</sup>, 2017.

**1.5 Objectives** Using lay language, describe the purpose, specific aims, or objectives that will be met by this specific project. If hypotheses are being tested, describe them. You will be asked to describe the specific procedures in a later section.

If your application involves the use of a HUD "humanitarian" device: describe whether the use is for "on-label" clinical patient care, "off-label" clinical patient care, and/or research (collecting safety and/or effectiveness data).

Orthodontic tooth movement induces an inflammatory response that can cause patients mild to moderate pain, especially within the first few days after forces have been applied. It has been shown that the use of over-the-counter analgesics such as acetaminophen and NSAIDs (i.e. ibuprofen) can be used effectively in the treatment of mild to moderate pain caused by orthodontic tooth movement. When such analgesics are taken preemptively to the introduction of orthodontic forces, a greater reduction in postoperative pain has been reported.

The combined use of acetaminophen and ibuprofen has been shown to have an additive relationship in the control of mild to moderate dental pain following tooth extractions. While each drug can individually reduce pain, the combination has been shown to be even more efficacious.

This study is designed to determine if the preemptive use of a combination of acetaminophen and ibuprofen is more effective in reducing dental pain following orthodontic treatment when compared to the use of acetaminophen and ibuprofen alone.

### Hypothesis:

Patients taking a combination of acetaminophen and ibuprofen prior to orthodontic treatment will report less pain when compared to those that premedicate with acetaminophen or ibuprofen alone.

(1.6) Study design. Provide a one-sentence description of the general study design and/or type of methodology.

Your answer will help HSD in assigning applications to reviewers and in managing workload. Examples: a longitudinal observational study; a double-blind, placebo-controlled randomized study; ethnographic interviews; web scraping from a convenience sample of blogs; medical record review; coordinating center for a multi-site study.

Double-blind randomized control study

1.7 Intent. Check all the descriptors that apply to your activity. You must place an "X" in at least one box.

This question is essential for ensuring that your application is correctly reviewed. Please read each option carefully.

| Descriptor |
|---|
| 1. Class project or other activity whose purpose is to provide an educational experience for the researcher (for example, to learn about the process or methods of doing research). |
| 2. Part of an institution, organization, or program's own internal operational monitoring. |
| 3. Improve the quality of service provided by a specific institution, organization, or program. |
| <ul> <li>4. Designed to expand the knowledge base of a scientific discipline or other scholarly field of study, and produce results that:</li> <li>Are expected to be applicable to a larger population beyond the site of data collection or the specific subjects studied, or</li> <li>Are intended to be used to develop, test, or support theories, principles, and statements of relationships, or to inform policy beyond the study.</li> </ul> |
| 5. Develop information about a drug or device through its prospective use and assignment to subjects, which will then be submitted to the Food and Drug Administration (FDA) in support of a marketing or research application for an investigational drug or device, or for changes to the purpose, population, or dose for an already-approved drug or device. |
| 6. Focus directly on the specific individuals about whom the information or biospecimens are collected through oral history, journalism, biography, or historical scholarship activities, to provide an accurate and evidence-based portrayal of the individuals. |
| 7. A quality improvement or program improvement activity conducted to improve the implementation (delivery or quality) of an accepted practice, or to collect data about the implementation of the practice for clinical, practical, or administrative purposes. This does not include the evaluation of the efficacy of different accepted practices, or a comparison of their efficacy. |
| 8. Public health surveillance activities conducted, requested, or authorized by a public health authority for the sole purpose of identifying or investigating potential public health signals or timely awareness and priority setting during a situation that threatens public health. |
| 9. Preliminary, exploratory, or research development activities (such as pilot and feasibility studies, or reliability/validation testing of a questionnaire) |
| 10. Expanded access use of a drug or device not yet approved for this purpose |
| 11. Use of a Humanitarian Use Device |
| 12. Other. Explain: |

- **1.8 Background, experience, and preliminary work**. Answer this question <u>only</u> if your proposed activity has one or more of the following characteristics. The purpose of this question is to provide the IRB with information that is relevant to its risk/benefit analysis.
  - Involves more than minimal risk (physical or non-physical)
  - Is a clinical trial, or
  - Involves having the subjects use a drug, biological, botanical, nutritional supplement, or medical device.

"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests.

**a.** <u>Background</u>. Provide the rationale and the scientific or scholarly background for your proposed activity, based on existing literature (or clinical knowledge). Describe the gaps in current knowledge that your project is intended to address.

Do not provide scholarly citations. Limit your answer to less than one page, or refer to an attached document with background information that is no more than three pages long.

Pain associated with orthodontic tooth movement is generated by an inflammatory process. This hyperalgesic result can reduce patient compliance and may be a deterrent for treatment for some individuals. Prostaglandins are one of the primary mediators of this inflammatory response and are synthesized by the enzyme cyclooxygenase (COX), which exists as two forms: COX-1 (constitutive), and COX-2 (inducible). The use of non-steroidal anti-inflammatory drugs (NSAIDs) have been shown to inhibit the activity of COX, thus achieving some of its analgesic effect by its anti-inflammatory properties.<sup>1</sup>

Numerous studies have shown the use of analgesics, such as NSAIDs and acetaminophen, to be effective in the control and management of pain induced by orthodontic tooth movement.<sup>2, 3, 4</sup> Preemptive administration of analgesics an hour before the placement of orthodontic separators has been shown to have a greater reduction in pain than analgesic administration following the procedure.<sup>5, 6, 7</sup> Acetaminophen (650mg) and ibuprofen (400mg) have been shown to be similarly effective as a pre-emptive analgesic for the control of dental pain following separator and initial archwire placement.<sup>4, 8, 9</sup>

The combined use of acetaminophen and ibuprofen has been demonstrated to be more effective than either medication alone for the treatment of post-operative dental pain. The combination of acetaminophen with NSAIDs has been shown to have a synergistic relationship in reducing visceral pain in a rat model. It has been suggested that the simultaneous use acetaminophen and NSAIDs has held an additive analgesic effect against other prostaglandin mediated pain such as osteoarthritis, dental surgery, and other surgical procedures. It

To our knowledge, there is no research that has been done that investigates the pre-emptive use of a combination of acetaminophen and ibuprofen for the control of dental pain associated with orthodontic treatment. We are interested in discovering if the recommended use of a combination of analgesics for the control of dental pain can be used pre-emptively in the orthodontic setting.

#### References:

- 1. Krishnan V; Orthodontic pain: from causes to management—a review. Eur J Orthod 2007; 29 (2): 170-179. doi: 10.1093/ejo/cjl081.
- 2. Sudhakar V, Vinodhini T S, Mohan A M, Srinivasan B, Rajkumar B K. The efficacy of different pre- and post-operative analgesics in the management of pain after orthodontic separator placement: A randomized clinical trial. J Pharm Bioall Sci 2014;6, Suppl S1:80-4.
- 3. Simmons KE, Brandt M. Control of orthodontic pain. Journal of the Indiana Dental Association, 1992, vol. 71 (pg. 8-10).
- 4. Ngan P, Wilson S, Shanfeld J, Amini H. The effect of ibuprofen on the level of discomfort in patients undergoing orthodontic treatment. American Journal of Orthodontics and Dentofacial

Orthopedics, 1994, vol. 106 (pg. 88-95).

- 5. Steen Law SL, Southard KA, Law AS, Logan HL, Jakobsen JR. An evaluation of preoperative ibuprofen for treatment of pain associated with orthodontic separator placement. *American Journal of Orthodontics and Dentofacial Orthopedics*, 2000, vol. 118 (pg. 629-633).
- 6. Bernhardt MK, Southard KA, Batterson KD, Logan HL, Baker KA, Jakobsen JR. The effect of preemptive and/or postoperative ibuprofen therapy for orthodontic pain. *American Journal of Orthodontics and Dentofacial Orthopedics*, 2001, vol. 120 (pg. 20-27).
- 7. Polat O, Kararam AI, Durmus E. Effects of preoperative ibuprofen and naproxan sodium on orthodontic pain. The Angle Orthodontist, 2005, vol. 75 (pg. 791-796).
- 8. Zarif Najafi H, Oshagh M, Salehi P, Babanouri N, Torkan S. Comparison of the effects of preemptive acetaminophen, ibuprofen, and meloxicam on pain after separator placement: a randomized clinical trial. *Progress in Orthodontics*. 2015;16:34. doi:10.1186/s40510-015-0104-y.
- 9. Bird S, Williams K, Kula K. Preoperative acetaminophen vs ibuprofen for control of pain after orthodontic separator placement. Am J Ortho Dentofacial Orthop. 2007;132:504–10. doi: 10.1016/j.aiodo.2006.11.019
- 10. Merry AF, Gibbs RD, Edwards J, et al. Combined acetaminophen and ibuprofen for pain relief after oral surgery in adults: a randomized controlled trial. *BJA: British Journal of Anaesthesia*. 2010;104(1):80-88. doi:10.1093/bja/aep338.
- 11. Bailey E, Worthington HV, van Wijk A, Yates JM, Coulthard P, Afzal Z. Ibuprofen and/or paracetamol (acetaminophen) for pain relief after surgical removal of lower wisdom teeth. Cochrane Database Svst Rev. 2013 Dec 12:(12):CD004624. doi:10.1002/14651858.CD004624.pub2.
- 12. Moore PA, Hersh EV. Combining ibuprofen and acetaminophen for acute pain management after third-molar extractions: translating clinical research to dental practice. *Journal of American Dental Association*. 2013 Aug;144(8):898-908.
- 13. Miranda HF, Puig MM, Prieto JC, Pinardi G. Synergism between paracetamol and nonsteroidal anti-inflammatory drugs in experimental acute pain. Pain. 2006 Mar;121(1-2):22-8. Epub 2006 Feb 9. doi: 10.1016/j.pain.2005.11.012.
  - 14. Altman RD. A rationale for combining acetaminophen and NSAIDs for mild-to-moderate pain. Clinical and Experimental Reumatology, 22 (2004), pp. 110–117.
- **b.** Experience and preliminary work. Briefly describe experience or preliminary work or data (if any) that you or your team have that supports the feasibility and/or safety of this study.

It is not necessary to summarize all discussion that has led to the development of the study protocol. The IRB is interested only in short summaries about experiences or preliminary work that suggest the study is feasible and that risks are reasonable relative to the benefits. Examples: You have already conducted a Phase 1 study of an experimental drug which supports the Phase 2 study you are now proposing to do; you have already done a small pilot study showing that the reading skills intervention you plan to use is feasible in an after-school program with classroom aides; you have experience with the type of surgery that is required to implant the study device; you have a study coordinator who is experienced in working with subjects who have significant cognitive impairment.

The Orthodontics Graduate Clinic currently recommends the use of analgesics for pain management.

**1.9 Supplements**. Check all boxes that apply, to identify Supplements you should complete and upload to the **Supporting Documents** SmartForm in **Zipline**.

This section is here instead of at the end of the form to reduce the risk of duplicating information in this IRB Protocol form that you will need to provide in these Supplements.

| Check all<br>That Apply | Type of Research | Supplement Name |
|---|---|---|
| | <b>Department of Defense</b> The research involves Department of Defense funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Defense |
| | Department of Energy The research involves Department of Energy funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Energy |
| x | <b>Drug, biologic, botanical, supplement</b> Procedures involve the use of <u>any</u> drug, biologic, botanical or supplement, even if the item is not the focus of your research | ZIPLINE SUPPLEMENT:<br>Drugs |
| | Emergency exception to informed consent Research that requires this special consent waiver for research involving more than minimal risk | ZIPLINE SUPPLEMENT: Exception from Informed Consent for Emergency Research (EFIC) |

| Include: -Age 12-5 Exclude p -History o -Hyperser -Aspirin-s -Renal or -History o -Cardiova -Currently -Bleeding -Pregnant 2.3 Prisoners. intended ta a. Will you | patient with: of taking an analgesic in the past six hours institutive to ibuprofen or acetaminophen sensitive asthma liver impairment of GI bleeding or ulcers ascular disease, recent myocardial infarction, heart failure, or coronary artery by y taking antibiotics or other medications for a chronic systemic disease g disorder to or nursing IRB approval is required in order to include prisoners in research, even when p arget population. recruit or obtain data from individuals that you know to be prisoners? Individuals that you know to be prisoners are not a target worksheet: Prisoners for the definition of "prisoner". | pass graft surgery<br>risoners are not an |
|---|---|---|
| Include: -Age 12-5 Exclude p -History o -Hyperser -Aspirin-s -Renal or -History o -Cardiova -Currently -Bleeding -Pregnant 2.3 Prisoners. intended ta a. Will you | patient with: of taking an analgesic in the past six hours institutive to ibuprofen or acetaminophen sensitive asthma liver impairment of GI bleeding or ulcers ascular disease, recent myocardial infarction, heart failure, or coronary artery by y taking antibiotics or other medications for a chronic systemic disease g disorder t or nursing IRB approval is required in order to include prisoners in research, even when p arget population. recruit or obtain data from individuals that you know to be prisoners? Individuals that you know to be prisoners are not a target | pass graft surgery<br>risoners are not an |
| Exclude programmer - Age 12-5 Exclude programmer - History or - History or - Cardiovar - Currently - Bleeding - Pregnant 2.3 Prisoners intended to | patient with: of taking an analgesic in the past six hours institutive to ibuprofen or acetaminophen sensitive asthma liver impairment of GI bleeding or ulcers ascular disease, recent myocardial infarction, heart failure, or coronary artery by ye taking antibiotics or other medications for a chronic systemic disease gedisorder to or nursing IRB approval is required in order to include prisoners in research, even when parget population. | pass graft surgery |
| Exclude programmer of the study from Include: -Age 12-5 Exclude programmer of the study of the | patient with: of taking an analgesic in the past six hours insitivity to ibuprofen or acetaminophen sensitive asthma liver impairment of GI bleeding or ulcers ascular disease, recent myocardial infarction, heart failure, or coronary artery by y taking antibiotics or other medications for a chronic systemic disease g disorder to or nursing | pass graft surgery |
| | t among interested or potential subjects. Define any technical terms in lay langu | uage. |
| | nd exclusion criteria. Describe the specific criteria you will use to decide who v | |
| gender, he | ts. Describe the general characteristics of the subject populations or groups, included the status, and any other relevant characteristics. d females aged 12-59 in good health currently in orthodontic treatment. | cluding age range, |
| 2 PARTICIPA | | 1 10 |
| | · <u> </u> | |
| | None of the above | |
| | Participant results sharing Individual research results will be shared with subjects. | ZIPLINE SUPPLEMENT: Participant Results Sharing |
| | Multi-site study (You are asking the UW IRB to review one or more sites in a multi-site study.) | ZIPLINE SUPPLEMENT: Participating Site in Multi- Site Research |
| | Medical device Procedures involve the use of <u>any</u> medical device, even if the device is not the focus of your research, except when the device is FDA-approved and is being used through a clinical facility in the manner for which it is approved | ZIPLINE SUPPLEMENT: Devices |
| | | Genomic Data Sharing |
| | Genomic data sharing Genomic data are being collected and will be deposited in an external database (such as the NIH dbGaP database) for sharing with other researchers | ZIPLINE SUPPLEMENT: |

Version 1.3

| • | <ul> <li>Yes → If yes, answer the following questions (i – iv).</li> <li>i. Describe the type of prisoners, and which prisons/jails:</li> </ul> |
|---|---|
| general living cond<br>earnings in prison | t prisoner research is whether the effect of participation on prisoners' litions, medical care, quality of food, amenities, and opportunity for will be so great that it will make it difficult for prisoners to adequately rch risks. What will you do to reduce the chances of this? |
| procedures will be | iii. Describe what you will do to make sure that (a) your recruitment and subject selection<br>procedures will be fair to all eligible prisoners and (b) prison authorities or other prisoners will<br>not be able to arbitrarily prevent or require particular prisoners from participating. |
| Washington State<br>encourage or facil<br>decisions, and (b) | iv. If your research will involve prisoners in federal facilities or in state/local facilities outside of Washington State: check the box below to provide your assurance that you will (a) not encourage or facilitate the use of a prisoner's participation in the research to influence parole decisions, and (b) clearly inform each prisoner in advance (for example, in a consent form) that participation in the research will have no effect on his or her parole. |
| Confirmed | |
| <b>b.</b> Is your research likely to have subj | ects who become prisoners while participating in your study? |
| For example, a longitudinal study of y point during the study. | outh with drug problems is likely to have subjects who will be prisoners at some |
| <b>—</b> | s, describe the procedures and/or data collection you will continue with oner subjects |
| <b>2.4 Protected populations</b> . IRB approval is required for the use of the subject populations listed here. Check the boxes for any of these populations that you will purposefully include in your research. (In other words, being a part of the population is an inclusion criterion for your study.) | |
| Population | approval but do not need to be completed or submitted. Worksheet |
| Children | <u>WORKSHEET: Children</u><br> |
| Children who are wards | WORKSHEET: Children |
| Fetuses in utero | WORKSHEET: Pregnant Women |
| Neonates of uncertain viability | WORKSHEET: Neonates |
| Version 1.3 ZIPLINE APPLICATION: IRB Protocol #2003 | |

| No | n-viable neonates | WORKSHEET: Neonates |
|---|---|---|
| Pre | egnant women | WORKSHEET: Pregnant Women |
| | arch and its specific setting. This will vary according | the legal age for consent to treatments or procedures involved in to the location of the research (that is, for different states and |
| • | check any of the boxes above, use this space t<br>RB to consider. | o provide any information you think may be relevant for |
| | | . Will you actively recruit from Native American or non-U.S. organization, or similar community-based organization? |
| | particular territory and their cultural or historical dis | gislation as having a set of specific rights based on their historical stinctiveness from other populations that are often politically |
| Example | s: a reservation school or health clinic; recruiting du | ring a tribal community gathering |
| X No | → If yes, name the tribe, tribal-focused org | ganization, or similar community based organization. The al/indigenous approval before beginning your research. |
| Commo | | le information about other individuals from your subjects? information or contact information about family members, |
| your rese<br>your sub | earch team to <u>readily identify</u> the person. For examp<br>jects several questions about their grandparents but | one or in combination, would allow you or another member of the, suppose that you are studying immigration history. If you ask to you do not obtain names or other information that would allow llecting private identifiable information about the grandparents. |
| X No | | I human subjects in your study. Describe them and what |
| | r <b>of subjects.</b> Can you predict or describe the m<br>te your study, for each subject group? | naximum number of subjects (or subject units) you need to |
| interest i | units mean units within a group. For most research s<br>in some research is not the individual. Examples:<br>Dyads such as caregiver-and-Alzheimer's patient, or<br>Families<br>Other units, such as student-parent-teacher | tudies, a group will consist of individuals. However, the unit of |

#2003

<u>Subject group</u> means categories of subjects that are meaningful for your research. Some research has only one subject group – for example, all UW students taking Introductory Psychology. Some common ways in which subjects are grouped include:

- By intervention for example, an intervention group and a control group.
- By subject population or setting for example, urban versus rural families
- By age for example, children who are 6, 10, or 14 years old.

The IRB reviews the number of subjects you plan to study in the context of risks and benefits. You may submit a Modification to increase this number at any time after you receive IRB approval. If the IRB determines that your research involves no more than minimal risk: you may exceed the approved number and it will not be considered non-compliance. If your research involves more than minimal risk: exceeding the approved number will be considered non-compliance.

No

→ If no, provide your rationale in the box below. Also, provide any information you can about the scope/size of the research. You do not need to complete the table.

Example: you may not be able to predict the number of subjects who will complete an online survey advertised through Craigslist, but you can state that you will post your survey for two weeks and the number who respond is the number who will be in your study.

X Yes

→ If yes, for each subject group, use the table below to provide your estimate of the maximum desired number of individuals (or other subject unit, such as families) who will complete the research.

| Group name/description | Maximum desired number of individuals (or other subject unit, such as families) who will complete the research *For clinical trials: provide numbers for your site and for the study-wide total number |
|---|---|
| Acetaminophen/Ibuprofen | 60 |
| Acetaminophen | 60 |
| Ibuprofen | 60 |

### **3 INTERNATIONAL RESEARCH SETTING**

Answer the questions in this section ONLY if your research will occur at sites outside of the United States

**3.1 Reason for sites**. Describe the reason(s) why you selected the sites where you will conduct the research.

**3.2 Local context**. Culturally-appropriate procedures and an understanding of local context are an important part of protecting subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect your research or how it is conducted.

Examples: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male researcher; instead, the researcher may need to ask a male family member for permission before the woman can be approached. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual members of a group.

This federal site maintains an international list of human research standards and requirements: <a href="http://www.hhs.gov/ohrp/international/index.html">http://www.hhs.gov/ohrp/international/index.html</a>

|----------|
| D 44 C20 |

- **3.3 Site-specific laws**. Describe any local laws that may affect your research (especially the research design and consent procedures). The most common examples are laws about:
  - **Specimens** for example, some countries will not allow biospecimens to be taken out of the country.
  - Age of consent laws about when an individual is considered old enough to be able to provide consent vary across states, and across countries.
  - **Legally authorized representative** laws about who can serve as a legally authorized representative (and who has priority when more than one person is available) vary across states and countries.
  - **Use of healthcare records** many states (including Washington State) have laws that are similar to the federal HIPAA law but that have additional requirements.

| 3.4 Site-specific administrative or ethical requirements. | Describe local administrative or ethical requirements that |
|---|---|
| affect your research. | |

Example: A school district may require you to obtain permission from the head district office as well as school principals before approaching teachers or students; a factory in China may allow you to interview factory workers but not allow you to pay them.

### **4 RECRUITING and SCREENING PARTICIPANTS**

**4.1** Recruiting and Screening. Describe how you will identify, recruit, and screen subjects. Include information about: how, when, where, and in what setting. Identify who (by position or role, not name) will approach and recruit subjects, and who will screen them for eligibility.

Patients of the University of Washington Department of Orthodontics that are scheduled for archwire adjustments from March to June 2017 will be screened for this study. Upon check in for their appointment, the clinic will be instructed to provide the patient with a recruitment flyer regarding the study. Interested participants will return the flyer to the front desk and the principal investigator will meet with them before the scheduled appointment to review the consent form. Participants will be asked if they meet all of the eligibility requirements that are outlined on the application. The consent form will have a description of the study included in it and will be used to help answer any questions that the participant may have.

#### 4.2 Recruitment materials.

a. What materials (if any) will you use to recruit and screen subjects?

Examples: talking points for phone or in-person conversations; video or audio presentations; websites; social media messages; written materials such as letters, flyers for posting, brochures, or printed advertisements; questionnaires filled out by potential subjects.

Recruitment flyers will be available for the front office staff of the clinic. The front office staff is able to view the reason for the appointment and will distribute the recruitment flyer when the patient checks in. The consent form will be used to help explain the details of the study as well as answer any questions.

|-------|
| _ |

**b.** Upload descriptions of each type of material (or the materials themselves) to the **Consent Forms and Recruitment Materials** SmartForm of **Zipline**. If you will send letters to the subjects, the letter should include a statement about how you obtained the subject's name, contact information, and any other subject-specific information (such as a health condition) that is mentioned in the letter.

HSD encourages researchers to consider uploading descriptions of most recruitment and screening materials instead of the materials themselves. The goal is to provide the researchers with the flexibility to change some information on the materials without submitting a Modification for IRB approval of the changes. Examples:

- You could provide a list of talking points that will be used for phone or in-person conversations instead of a script.
- For the description of a flyer, you might include the information that it will provide the study phone number and the name of a study contact person (without providing the actual phone number or name). In doing so, you would not need to submit a Modification if/when the study phone number or contact person changes. Also, instead of listing the inclusion/exclusion criteria, you might state that the flyer will list one or a few of the major inclusion/exclusion criteria.
- For the description of a video or a website, you might include a description of the possible visual elements and a list of the content (e.g., study phone number; study contact person; top three inclusion/exclusion criteria; payment of \$50; study name; UW researcher).
- **4.3 Relationship with participant population**. Do any members of the study team have an existing relationship with the study population(s)?

Examples: a study team member may have a dual role with the study population (for example, being their clinical care provider, teacher, laboratory directory or tribal leader in addition to recruiting them for his/her research).



→ If yes, describe the nature of the relationship.

- **4.4 Payment to participants**. Describe any payment you will provide, including:
  - The total amount/value
  - Whether payment will be "pro-rated" so that participants who are unable to complete the research may still receive some part of the payment

The IRB expects the consent process or study information provided to the subjects to include information about the number and amount of payments, and especially the time when subjects can expect to receive payment. One of the most frequent complaints received by HSD is from subjects who expected to receive cash or a check on the day that they completed a study and who were angry or disappointed when payment took 6-8 weeks to reach them.

Do not include a description of any expenses that will be reimbursed.

When the participants return the completed workbook they will be able to enter a raffle for one of four \$50 VISA gift cards. The participant will tear off the provided card on last page of their workbook, write their contact information, and place it in a locked collection box. Participants that elected to complete the electronic version of the workbook will be entered into the raffle when their last entry has been submitted. At the conclusion of the study, four of the raffle tickets will be randomly drawn. The winners will be contacted and instructed to claim their prize at the front office at their next appointment or at an agreed upon time.

ZIPLINE APPLICATION: IRB Protocol

| #2003 |
|-------|

| <b>1.5 Non-monetary compensation</b> . Describe any non-monetary compensation you will provide. Example: extra credit for students; a toy for a child. If you will be offering class credit to students, you must provide (and describe) an alternate way for the students to earn the extra credit without participating in your research. |
|---|
| 6.6 Consent for recruiting and screening. Will you obtain consent for any of the recruiting and screening procedures (Section 8: Consent of Adults asks about consent for the main study procedures). |
| "Consent" includes: consent from individuals for their own participation; parental permission; assent from children; consent from a legally authorized representative for adult individuals who are unable to provide consent. |
| <ul> <li>Examples:</li> <li>For a study in which names and contact information will be obtained from a registry: the registry should have conse from the registry participants to release their names and contact information to researchers.</li> <li>For a study in which possible subjects are identified by screening records: there will be no consent process.</li> <li>For a study in which individuals respond to an announcement and call into a study phone line: the study team personalizing to the individual may obtain non-written consent to ask eligibility questions over the phone.</li> </ul> |
| X No → If no, you must still answer <u>question 4.7</u> below. |
| Yes → If yes, describe the consent process. |
| <ul> <li>a. <u>Documentation of consent</u>. Will you obtain a written or verifiable electronic signature from the subject on a consent form to document consent for all of the <u>recruiting and screening procedures</u>?</li> <li>No</li> <li>If no, describe the information you will provide during the consent process and for which procedures.</li> </ul> |
| Yes → If yes, upload the consent form to the Consent Forms and Recruitment Materia |
| page of <b>Zipline</b> . |
| .7) Data and specimens for recruiting and screening. For studies where you will obtain consent, describe any data and/or specimens (including any PHI) you will obtain for recruiting and screening (prior to obtaining consent) and whether you will retain it as part of the study data. |
| <b>Obtain</b> means to possess or record in any fashion (writing, electronic document, video, email, voice recording, etc.) for research purposes and to retain for any length of time. |
| Examples: names and contact information; the information gathered from records that were screened; results of screening questionnaires or screening blood tests; Protected Health Information (PHI) from screening medical records to identify possible subjects. |
| The front office staff that will be distributing the recruitment flyers will not obtain any additional data from this study than they normally would. The research team will not obtain any data until the participant has expressed interest. |
| ZIPLINE APPLICATION: IRB Protocol #20 |

### **5 PROCEDURES**

5.1) Study procedures. Using lay language, provide a complete description of the study procedures, including the sequence, intervention or manipulation (if any), time required, and setting/location. If it is available and you think it would be helpful to the IRB: Upload a study flow sheet or table to the Supporting Documents SmartForm in Zipline.

<u>For studies comparing standards of care</u>: It is important to accurately identify the research procedures. See UW IRB <u>POLICY</u>:
<u>Risks of Harm from Standard Care</u> and the draft guidance from the federal Office of Human Research Protections, <u>"Guidance on Disclosing Reasonably Foreseeable Risks in Research Evaluating Standards of Care"</u>; October 20, 2014.

There will be three groups of medication: acetaminophen (650mg); ibuprofen (400mg); and acetaminophen (650mg) + ibuprofen (400mg). The medications will be prepared by the Kelley-Ross Compounding Group (Seattle, WA) to make each medication similar in appearance in order to prevent recognition of the medication by the investigator or participant. The medications will be placed in individual vials and labeled as either A, B, or C. A sealed document will be sent with the medications that can properly identify which medications were assigned to each group, and this document will not be opened until the conclusion of the study.

During the informed consent process, participants will be asked if they meet all of the eligibility requirements that are outlined on the recruitment flyer. After reviewing and signing the informed consent, each eligible patient will be given a workbook that has a pre-designated participant number. A master list will be made in Microsoft Excel that uses a random number generator to randomly assign each participant number to Group A, B, or C, which will correspond to the indicated medication that is to be delivered. The appropriate medication will be administered with a 3 oz. paper cup of water. The patient will give the provider the first page of the workbook to complete. The provider will record the patient' age, gender, and give a brief description of the treatment that will be completed at the appointment. Once completed, the information will be returned to the principal investigator at the front desk.

Pain intensity will be measured using a numerical visual analog scale (VAS) immediately following drug administration, 6 hours after orthodontic treatment, the next morning after orthodontic treatment, the second morning after orthodontic treatment. At the aforementioned time periods, the participant will record their pain on the VAS for each of the following scenarios: teeth at rest, back teeth lightly touching, and when chewing a small piece (~0.5 inch) of provided wax. Participants will be instructed to not use other analgesics during the week if they can help it. If the participant must use an analgesic, they should record the time, name, and amount taken.

The participant will have the option to complete the recordings digitally through the website Catalyst. If the participant does not wish to complete the submissions online, then they will be given paper copies of the workbook to take home with them. Once completed, the patient can return the workbook at their next appointment. When returning the completed workbook, participants have the option of tearing off the last page of their workbook, writing their contact information, and entering it into a raffle for one of four \$50 gift cards. Participants electing to complete the recordings digitally will be entered into the raffle upon submission of their last recording.

The recordings from the VAS workbooks will becompiled in Microsoft Excel.

There will be three groups of medication: acetaminophen (650mg); ibuprofen (400mg); and acetaminophen (650mg) + ibuprofen (400mg). The medications will be prepared by the Kelley-Ross Compounding Group (Seattle, WA) to make each medication similar in appearance in order to prevent recognition of the medication by the investigator or participant. The medications will be placed in individual vials and labeled as either A, B, or C. A sealed document will be sent with the medications that can properly identify which medications were assigned to each group, and this document will not be opened until the conclusion of the study.

During the informed consent process, participants will be asked if they meet all of the eligibility requirements that are outlined on the recruitment flyer. After reviewing and signing the informed consent, each eligible patient will be given a workbook that has a pre-designated participant number. A master list will be made in Microsoft Excel that uses a random number generator to randomly assign each participant number to Group A, B, or C, which will correspond to the indicated medication that is to


be delivered. The appropriate medication will be administered with a 3 oz. paper cup of water. The patient will give the provider the first page of the workbook to complete. The provider will record the patient' age, gender, and give a brief description of the treatment that will be completed at the appointment. Once completed, the information will be returned to the principal investigator at the front desk.

Pain intensity will be measured using a numerical visual analog scale (VAS) immediately following drug administration, 6 hours after orthodontic treatment, the next morning after orthodontic treatment, the second morning after orthodontic treatment. At the aforementioned time periods, the participant will record their pain on the VAS for each of the following scenarios: teeth at rest, back teeth lightly touching, and when chewing a small piece (~0.5 inch) of provided wax. Participants will be instructed to not use other analgesics during the week if they can help it. If the participant must use an analgesic, they should record the time, name, and amount taken.

The participant will have the option to complete the recordings digitally through the website Catalyst. If the participant does not wish to complete the submissions online, then they will be given paper copies of the workbook to take home with them. Once completed, the patient can return the workbook at their next appointment. When returning the completed workbook, participants have the option of tearing off the last page of their workbook, writing their contact information, and entering it into a raffle for one of four \$50 gift cards. Participants electing to complete the recordings digitally will be entered into the raffle upon submission of their last recording.

The recordings from the VAS workbooks will be compiled in Microsoft Excel.

**5.2 Data variables.** Describe the specific data you will obtain (including a description of the most sensitive items). If you would prefer, you may upload a list of the data variables to the **Supporting Documents** SmartForm instead of describing the variables below.

Age, sex, description of treatment during the appointment, did the patient take any additional pain medications during the study, and pain scores during rest, light biting, and chewing at several time points (immediately following drug administration, 6 hours, the next morning, and the second morning after orthodontic treatment.

**(5.3) Data sources.** For all types of data that you will access or collect for this research: Identify whether you are obtaining the data from the subjects (or subjects' specimens) or whether you are obtaining the data from some other source (and identify the source).

If you have already provided this information in Question 5.1, you do not need to repeat the information here.

Patient appointments for the University of Washington Department of Orthodontics clinic during March to June 2017 will be screened for arch wire adjustment appointments. The applicable appointments will be given a recruitment flyer.

Patients will be given a paper or online workbook to record their pain on a visual analogue scale (VAS) to return at their next scheduled appointment and their provider will complete a short questionnaire.

- **5.4 Retrospective/prospective.** For all types of data and specimens that you will access or collect for this research: Describe which data are:
  - Retrospective (i.e., exist at the time when you submit this application)
  - Prospective (i.e., do not yet exist at the time when you submit this application)
  - Both retrospective and prospective (for example, past and future school records)

| Prospective: | Workbook of | f pain | record | ings and | d quest | ionnair |
|--------------|--------------|--------|--------|----------|---------|---------|
| Both: Patien | t appointmen | ts for | archwi | re adius | tments | |

| #2003 |
|-------|

**5.5 Identifiability of data and specimens**. Answer these questions carefully and completely. This will allow HSD to accurately determine the type of review that is required and to assist you in identifying relevant compliance requirements. Review the following definitions before answering the questions:

Access means to view or perceive data, but not to possess or record it. See, in contrast, the definition of "obtain". Identifiable means that the identify of an individual is or may be readily (1) ascertained by the researcher or any other member of the study team from specific data variables or from a combination of data variables, or (2) associated with the information.

**Direct identifiers** are direct links between a subject and data/specimens. Examples include (but are not limited to): name, date of birth, medical record number, email or IP address, pathology or surgery accession number, student number, or a collection of your data that is (when taken together) identifiable.

**Indirect identifiers** are information that links between direct identifiers and data/specimens. Examples: a subject code or pseudonym.

**Key** refers to a single place where direct identifiers and indirect identifiers are linked together so that, for example, coded data can be identified as relating to a specific person. Example: a master list that contains the data code and the identifiers linked to the codes.

**Obtain** means to possess or record in any fashion (writing, electronic document, video, email, voice recording, etc.) for research purposes and to retain for any length of time. This is different from **accessing**, which means to view or perceive data.

| <b>a.</b> Will you or any n | nembers of your team have <u>access</u> to any direct or indirect identifiers? |
|---|---|
| Yes → | If yes, describe which identifiers and for which data/specimens. |
| | → If no, select the reason(s) why you (and all members of your team) will not have access to direct or indirect identifiers. |
| | X There will be no identifiers. |
| Ī | Identifiers or the key have been (or will have been) destroyed before you have access. |
| | You have (or will have) entered into an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to you under any circumstances. |
| _ | You should be able to produce this agreement for IRB upon request. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key to you. Describe them below. |
| _ | |
| <b>b.</b> Will you <u>obtain</u> a | ny direct or indirect identifiers? |
| $X$ Yes $\rightarrow$ | f yes, describe which identifiers and for which data/specimens. |
| _ | Participants may opt to sign up for text/email reminders to complete the recordings which would make it necessary for the research team to obtain the patient's phone number or email address. |
| _ | Patients may elect to be entered into a raffle at the end of their participation in the study. Participants can record their contact information on a blank card that will have no |

| | identifiers to their data. |
|---|---|
| | o, select the reason(s) why you (and all members of your team) will not obtain direct or irect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before you have access. |
| | You have (or will have) entered into an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to you under any circumstances. |
| | You should be able to produce this agreement for IRB upon request. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key to you. Describe them below. |
| <b>c.</b> If you obtain any ide | entifiers, indicate how the identifiers will be stored (and for which data). |
| | You will store the identifiers with the data. Describe the data to which this applies: |
| х | You will store identifiers and study data separately but you will maintain a link between the identifiers and the study data (for example, through the use of a code). Describe the data to which this applies: |
| | Participants electing to receive notifications to complete the submissions will have the provided contact information (phone number or email) recorded. The contact information will be recorded on a separate computer file than the data but linked with a participant number. |
| Х | You will store identifiers separately from the study data, with no link between the identifiers and the study data. Describe the data to which this applies: |
| | All data will be returned to the front office. There will be a locked box in the front office for participants to enter their contact information into. |
| research also collab<br>name of the collabo<br>Examples include but o | oration. Will individuals who provide you with coded information or specimens for your borate on other activities for this research? If yes, identify the activities and provide the orator's institution/organization. are not limited to: (1) study, interpretation, or analysis of the data that results from the coded thens; and (2) authorship on presentations or manuscripts related to this work. |
| , | |
| | ts. Will you use newborn dried bloodspots collected in the United States on or after |
| 1arch 18, 2015? | |
| X No | |
| n 1 3 | ZIPLINE APPLICATION: IRB Protocol #2003 |

| Ye s → | If yes, is this research supported by any federal funding (including any fellowship or career development award that provides salary support)? |
|---|---|
| | No Yes → If yes, describe how you will ensure that the bloodspots were collected with parental permission (in compliance with a 2015 law that applies to federal-funded research). |
| reason (for ex | alth Information (PHI). Will you access, obtain, use, or disclose a participant's identifiable PHI for any cample, to identify or screen potential subjects, to obtain study data or specimens, for study follownot involve the creation or obtaining of a Limited Data Set? |
| | ally-identifiable healthcare record information or clinical specimens from an organization considered a "covered ral HIPAA regulations, in any form or media, whether electronic, paper, or oral. |
| | If no, skip the rest of this question; go to question 5.8 If yes, answer all of the questions below. |
| | a. Describe the PHI you will access or obtain, and the reason for obtaining it. Be specific. |
| | Patient appointment information will be accessed for the UW-Orthodontics clinic for all patients for the duration of the study (April – June 2017) and will include name, phone number, and reason for visit. |
| | <ul> <li>b. Is any of the PHI located in Washington State?</li> <li>No</li> <li>X</li> <li>Yes</li> <li>c. Describe how you will access or obtain the PHI. Be specific.</li> </ul> |
| | When the patient checks-in for their appointment at the Orthodontics clinic, the front office staff members will be able to see the patient's name, phone number, and reason for their visit. If the reason for the visit for the patient involves archwire adjustment then the front office staff will hand the patient a recruitment flier. If the patient is interested in more information about participation in the study then the patient will notify the front office and will be greeted by the principal investigator. |
| | <b>d.</b> For which PHI will you obtain HIPAA authorization from the subjects by having them sign a HIPAA Authorization form, before obtaining and using the PHI? |
| | None |
| | Confirm by checking the box that you will use the UW Medicine HIPAA Authorization form maintained on the HSD website if you will access, obtain, use, or disclose UW Medicine PHI. Confirmed |
| | e. For which PHI will you NOT obtain HIPAA authorization from the subjects? |
| | Patient appointment information. |
| | Provide the following assurances by checking the boxes. The PHI will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research study, or for other research for which the use or |

| | disclosure of PHL would be permitted |
|---|---|
| | You will fulfill the HIPAA "accounting for disclosures" requirement. See UW Medicine Privacy Policy #25. THIS IS ONLY FOR UW RECORDS. |
| | There will be reasonable safeguards to protect against identifying, directly or indirectly, any patient in any report of the research. |
| | nta sharing. Will you obtain or generate genomic data (as defined at nih.gov/13faqs_gds.html)? |
| X No<br>Yes | → If yes, answer the question below. |
| _ | a. Is this research funded by NIH through a grant or contract application submitted to NIH on or after January 25, 2015? |
| | No Yes → If yes, you must comply with the NIH Genomic Data Sharing policy. Complete the <u>ZIPLINE SUPPLEMENT Genomic Data Sharing</u> and upload it to the Supporting Documents SmartForm of <i>Zipline</i> . |
| research us whether your only s Many federe data sharing data/specin | with other researchers or a repository/database, or to bank them for your own future unspecified es? You are strongly encouraged to consider the broadest possible future plans you might have, and u will obtain consent now from the subjects for future sharing or unspecified uses. Answer NO if naring will be through the NIH Genomic Data Sharing described in question 5.8. I grants and contracts now require data or specimen sharing as a condition of funding, and many journals require as a condition of publication. "Sharing" may include: informal arrangements to share your banked tens with other investigators; establishing a repository from which you formally share with others through written |
| _ | or sending your data/specimens to a third party repository/archive/entity such as the NIH dbGaP database, the e Open Access Repository (SSOAR), or the UCLA Ethnomusicology Archive. |
| s | <ul> <li>If yes, answer all of the questions below.</li> <li>a. Describe <u>what will be stored</u>, including whether any direct or indirect (e.g., subject codes) identifiers will be stored.</li> </ul> |
| | <b>b.</b> Describe what will be shared, including whether direct identifiers will be shared and (for specimens) what data will be released with the specimens. |
| | c. Who will oversee and/or manage the sharing?. |
| | <b>112222</b> |

| users. As stated above, consider the broadest possible uses. Examples: data will be used only for cardiovascular research; data w | vill not be used for research on |
|---|---|
| population origins. | mi not be useu joi research on |
| e. Consent. Will you obtain consent now from subjects for the b | anking and/or future sharing? |
| No | |
| Yes → If yes, be sure to include the information abo consent form (if there is one) and in your ans<br><u>Section 6</u> . | • |
| f. Withdrawal. Will subjects be able to withdraw their data/spe | cimens from banking or sharing? |
| No | |
| Yes → If yes, describe how, and whether there are a | • |
| Example: data can be withdrawn from the reposi<br>are released. | tory but cannot be retrieved after they |
| g. Agreements for sharing or release. Confirm by checking the (and, if applicable, UW Medicine) policies that require a form the recipient for release of data or specimens to individuals of databases. Data Use Agreements or Gatekeeping forms are used for data; Ma for specimens (or specimens plus data. Do not attach your template reviews nor approves them | al agreement between you and or entities other than federal terial Transfer Agreements are used |
| Confirmed | |
| <b>5.10 Communication with subjects during the study</b> . Describe the types of commu already-enrolled subjects during the study. Provide a description instead of the | |
| Examples: email, texts, phone, or letter reminders about appointments or about returning questionnaire; requests to confirm contact information. | ng study materials such as a |
| If requested, participants will receive email or text message notifications as resubmissions. | ninders to complete the |
| <b>5.11 Future contact with subjects</b> . Do you plan to retain any contact information you they can be contacted in the future? No | ou obtain for your subjects so that |
| Yes → If yes, describe the purpose of the future contact, and whether upon be limited to your team; if not, describe who else could be provided be provided by the provided by the provided provided by the p | ded with the contact information. |
| Examples: inform subjects about other studies; ask subjects for addition access that is not currently part of the study proposed in this application | - |
| Upon completion of the study, the participant will write the ticket and drop it into a locked box at the front desk of the drawn at the conclusion of the study and the respective indi | elinic. Four raffle tickets will be |

**d.** Describe the possible future uses, including limitations or restrictions (if any) on future uses or

notified to claim their prize at the front desk at a convenient time or their next appointment. All raffle tickets will be destroyed.

**5.12 Alternatives to participation.** Are there any alternative procedures or treatments that might be advantageous to the subjects?

If there are no alternative procedures or treatments, select "No". Examples of advantageous alternatives: earning extra class credit in some time-equivalent way other than research participation; obtaining supportive care or a standard clinical treatment from a health care provider instead of participating in research with an experimental drug.

| No |
|----|
| Va |

Yes → If yes, describe the alternatives.

- 5.13 Upload to the Supporting Documents SmartForm of Zipline all data collection forms (if any) that will be directly used by or with the subjects, and any scripts/talking points you will use to collect the data. Do not include data collection forms that will be used to abstract data from other sources (such as medical or academic records, or video recordings.
  - **Examples**: survey, questionnaires, subject logs or diaries, focus group questions.
  - **NOTE:** Sometimes the IRB can approve the general content of surveys and other data collection instruments rather than the specific form itself. This prevents the need to submit a modification request for future minor changes that do not add new topics or increase the sensitivity of the questions. To request this general approval, use the text box below to identify the questionnaires/surveys/ etc. for which you are seeking this more general approval. Then briefly describe the scope of the topics you will cover and the most personal and sensitive questions. The HSD staff person who screens this application will let you know whether this is sufficient or whether you will need to provide more information.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.
  - For data that will be gathered in an evolving way: This refers to data collection/questions that are not pre-determined but rather are shaped during interactions with participants in response to observations and responses made during those interactions. If this applies to your research, provide a description of the process by which you will establish the data collection/questions as you interact with subjects, how you will document your data collection/questions, the topics you plan to address, the most sensitive type of information you will plan to gather, and the limitations (if any) on topics you will raise or pursue.

Use this text box (if desired) to provide:

- Short written descriptions of materials that cannot be uploaded, such as URLs
- A description of the process you will use for data that will be gathered in an evolving way.
- The general content of questionnaires, surveys and similar instruments for which you are seeking general approval. (See the **NOTE** bullet point in the instructions above.)

The online version of the workbook is in the format of a Catalyst guiz. The online version asks for the participant number, the level of discomfort in the same three scenarios as the paper version of the workbook, and if the participant used any additional pain medications. All of the questions have an option of "I wish to skip this question."

https://catalyst.uw.edu/webg/survey/akeith/328766

5.14 Send HSD a Confidentiality Agreement if you will obtain or use any private identifiable UW records without subject's written consent (for example, screening medical records or class grades to identify possible subjects).

The Confidentiality Agreement form must be completed, printed, signed, and mailed to the Human Subjects Division at Box 359470. Your IRB application cannot be approved until we receive the Confidentiality Agreement.

|--------------------|
| -<br> |

## 6 CHILDREN (MINORS) and PARENTAL PERMISSION

**(6.1)Involvement of minors**. Does your research include minors (children)?

**Minor or child** means someone who has not yet attained the legal age for consent for the research procedures, as described in the applicable laws of the jurisdiction in which the research will be conducted. This may or may not be the same as the definition used by funding agencies such as the National Institutes of Health.

- In Washington State the generic age of consent is 18, meaning that anyone under the age of 18 is considered a child.
- There are some procedures for which the age of consent is much lower in Washington State. See the **WORKSHEET: Children** for details.

| • - | <ul> <li>The generic age of consent may be different in other states, and in other countries.</li> </ul> | | | | |
|---|---|---|---|---|---|
| No - | → If no, go to <u>Section 8</u> . | | | | |
| X Yes - | If yes, provide the age range of the nyour population(s). If there is more t | - | | ge for cons | ent in |
| | 12+ year old | | | | |
| Don't k | now true for some research invol | lving social | ne age of your subjects. For exam<br>media, the Internet, or a dataset<br>ernment agency. Go to <u>Section 8</u> | that you o | • |
| same as "pas<br>participate b<br>returned a fo | nission. Parental permission means ac<br>sive" or "opt out" permission where it<br>ecause they have been provided with in<br>rm indicating they don't want their chi | is assumed nformation | d that parents are allowing their on about the research and have no | children to | |
| <b>a.</b> Will you o | tain parental permission for: | | | | |
| All of y | our research procedures → Go | o to <mark>questi</mark> | on 6.2b. | | |
| None o | t volir research procedures | se the table<br>uestion 6.2 | e below to provide your justificati<br>b. | on, and ski | ip |
| Some of | Some of your research procedures Use the table below to identify the procedures for which you will not obtain written parental permission. | | | | |
| Be sure to con<br>specimens for | sider all research procedures and plans, inc<br>future work. | cluding scree | ening, future contact, and sharing/bo | anking of da | ta and |
| Children<br>Group <sup>1</sup> | Describe the procedures data/specimen collection (if a which there will be NO pare permission | any) for | Reason why you will not<br>obtain parental<br>permission | | u inform<br>bout the<br>arch? <sup>2</sup> |
| | | | | YES | NO |

ZIPLINE APPLICATION: IRB Protocol

Version 1.3


| | ĺ |
|---|---|
| | i — -<br>I |
| | i — -<br>I |
| | : <b>-</b> - |
| 1. If your answer is the same for all children groups or all procedures, you can collapse your answer across the groups and/or procedures. | |
| <ol> <li>Will you inform them about the research beforehand even though you are not obtaining active permission?</li> </ol> | |
| <b>b.</b> Indicate by checking the appropriate box(es) your plan for obtaining parental permission | |
| Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably available; or who only one parent has legal responsibility for the care and custody of the child | ŧη |
| One parent, even if the other parent is alive, known, competent, reasonably available, and shares legal responsibility for the care and custody of the child. | |
| This is all that is required for minimal risk research. | |
| If you checked both boxes, explain: | |
| Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advocate must be addition to any other individual acting on behalf of the child as guardian or in loco parentis. The same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). Your answer must address the following points: • Background and experience • Willingness to act in the best interests of the child for the duration of the research • Independence of the research, research team, and any guardian organization | in |
| 7 ASSENT OF CHILDREN (MINORS) | |
| Go to <u>Section 8</u> if your research does not involve children (minors). | |
| <b>7.1 Assent of children (minors)</b> . Though children do not have the legal capacity to "consent" to participate in research, they should be involved in the process if they are able to "assent" by having a study explained to them and/or by reading a simple form about the study, and then giving their verbal choice about whether they want t participate. They may also provide a written assent if they are older. See <a href="WORKSHEET: Children">WORKSHEET: Children</a> for circumstance in which a child's assent may be unnecessary or inappropriate. | 0 |
| a. Will you obtain assent for: | |
| X All of your research procedures and child groups → Go to question 7.2. | |
| None of your research procedures and child groups Use the table below to provide your justification, then skip to question 7.5. | |
| ZIPLINE APPLICATION: IRB Protocol #2 | .003 |

| Some of | your research procedures and child groups | → Use the table below to identify the procedures for which you will not obtain assent. |
|---|---|---|
| Be sure to consid<br>specimens for fu | | ning, future contact, and sharing/banking of data and |
| Children<br>Group¹ | Describe the procedures or data/specimen collection (if any) for which assent will NOT be obtained | Reason why you will not obtain assent |
| Table footnotes 1. If your answer is procedures. | the same for all children groups or all procedures, yo | ou can collapse your answer across the groups and/or |
| different ages, | | child group. If your research involves children of n are non-English speakers, include a description of u provide. |
| | | e study, I will read the assent form to the child and ild would like to continue, I will have them sign the |
| | stance. Describe how you will identify a child's of cations) during the research, and what you will | bjection or resistance to participation (including do in response. |
| If at any point no penalty. | the child does not wish to continue I will let the | m know that they are free to drop out of the study at |
| 7.4 Documentation assent? | of assent. Which of the following statements of | describes whether you will obtain documentation of |
| None of yo | our research procedures and child groups | → Use the table below to provide your justification, then go to question 7.4.a. |
| All of your | research procedures and child groups | → Go to question 7.4.a, do not complete the table |
| Some of y | our research procedures and/or child groups | → Complete the table below and then to go question 7.4.a |
| Children<br>Group <sup>1</sup> | Describe the procedures or data/specime collection (if any) for which assent will NOT be documented | n<br>Reason why you will not document assent |
| Version 1.3 | ZIPLINE APPLICATION: IRB Prot | #2003 |

#### Table footnotes

- 1. If your answer is the same for all children groups or all procedures, you can collapse your answer across the groups and/or procedures.
  - **a. Describe how you will document assent**. If the children are functionally illiterate or are not fluent in English, include a description of what you will do.

I will have the child sign the assent form.

- b. Upload all assent materials (talking points, videos, forms, etc.) to the Consent Form and Recruitment Materials SmartForm of *Zipline*. Assent materials are not required to provide all of the standard elements of adult consent; the information should be appropriate to the age, population, and research procedures. The documents should be in Word, if possible.
- 7.5 Children who reach the legal age of consent during participation in longitudinal research.

<u>Children who were enrolled at a young age and continue for many years</u>: It is best practice to re-obtain assent (or to obtain it for the first time, if you did not at the beginning of their participation).

<u>Children who reach the legal age of consent</u>: You must obtain informed consent from the now-adult subject for (1) any ongoing interactions or interventions with the subjects, or (2) the continued analysis of specimens or data for which the subject's identify is readily identifiable to the researcher, unless the IRB waives this requirement.

a. Describe your plans (if any) to re-obtain assent from children.

N/A

- b. Describe your plans (if any) to obtain consent for children who reach the legal age of consent.
  - If you plan to obtain consent, describe what you will do about now-adult subjects whom you are unable to contact.
  - If you do not plan to obtain consent or think that you will be unable to do so, explain why.

N/A

- **7.6 Other regulatory requirements**. (This is for your information only; no answer or response is required.)

  Researchers are responsible for determining whether their research conducted in schools, with student records, or over the Internet comply with permission, consent, and inspection requirements of the following federal regulations:
  - PPRA Protection of Pupil Rights Amendment
  - FERPA Family Education Rights and Privacy Act
  - COPPA Children's Online Privacy Protection Act

# **8 CONSENT OF ADULTS**

| eview the following definitions | before answering the questions in this section. |
|---|---|
| CONSENT | is the <u>process</u> of informing potential subjects about the research and asking them whether they want to participate. It usually (but not always) includes an opportunity for subjects to ask questions. It does not necessarily include the signing of a consent form. This question is about the consent process. |
| CONSENT DOCUMENTATION | refers to how a subject's decision to participate in the research is documented. This is typically obtained by having the subject sign a consent form. |

| CONSENT FORM | is a document signed by subjects, by which they a research as described in the consent form and in | |
|---|---|---|
| <b>ELEMENTS OF CONSENT</b> | ELEMENTS OF CONSENT are specific information that is required to be provided to subjects. | |
| PARENTAL PERMISSION | is the parent's active permission for the child to p<br>Parental permission is subject to the same require<br>written documentation of permission and require | ements as consent, including |
| SHORT FORM CONSENT | is an alternative way of obtaining written docume<br>commonly used with individuals who are illiterate<br>which translated consent forms are not available. | |
| WAIVER OF CONSENT | means there is IRB approval for not obtaining con the elements of consent in the consent process. | sent or for not including some of |
| WAIVER OF DOCUMENTATION OF CONSENT | means that there is IRB approval for not obtaining consent. | written documentation of |
| <b>8.1 Groups</b> Identify the groups to | which your answers in this section apply. | |
| Adult subjects Parents who are provided. | ing permission for their children to participate in re | |
| | NTS, the word "consent" below should also be inte | |
| permission and "sub<br>————————— | jects" should also be interpreted as applying to the | parents. |
| <b>8.2 The consent process</b> . This series of questions is about whether you will obtain consent for all procedures except recruiting and screening and, if yes, how. | | |
| The issue of consent for recruiting and screening activities is addressed in <u>question 4.6</u> . You do not need to repeat your answer to question 4.6. | | |
| <b>a</b> . Are there any procedures | or which you will not obtain consent? | |
| X No | | |
| • | the table below to identify the procedures for which acceptable answer for some studies. | h you will not obtain consent. |
| Be sure to consider all research parties for future work. | rocedures and plans, including future contact, and sharin | g/banking of data and specimens |
| Group <sup>1</sup> data/speci<br>any) for whi | he procedures or<br>men collection (if Reason why you will r<br>ch there will be NO consent<br>ent process | Will you<br>provide<br>not obtain subjects with<br>info about the<br>research after<br>they finish?<br>YES NO |

| <ul> <li>Table footnotes</li> <li>1. If your answer is the same for all groups you can collapse your answer across the groups and/or procedures</li> <li>b. Describe the consent process, if you will obtain consent for any or all procedures, for any or all groups and procedures separately if the consent processes are different.</li> </ul> | | ddress |
|---|---|---|
| Be sure to include: The location/setting where consent will be obtained Who will obtain consent (refer to positions, roles, or titles, not names). Whether/how you will provide an opportunity for questions How you will provide an adequate opportunity for the subjects to consider all options | or will see | oot the |
| When the subject returns the recruitment flyer to the check-in window, the principal investigat subject in the clinic's waiting area to review the elements of the study and answer any question | | eet the |
| c. <u>Comprehension</u> . Describe how you will ensure or test the subjects' understanding of the inforn consent process. | nation dui | ring the |
| After all questions are answered, the principal investigator will ask if the participant understanlike to continue with being a participant in the study. | ds and wo | ould |
| <b>d.</b> <u>Influence</u> . Does your research involve any subject groups that might find it difficult to say "no" because of the setting or their relationship with you, even if you don't pressure them to partici | | esearch |
| Examples: Student participants being recruited into their teacher's research; patients being recruited into provider's research, study team members who are participants; outpatients recruited from an outpatien room just prior to their surgery. | | |
| Yes → If yes, describe what you will do, for each of these subject groups, to reduce a setting or relationship on their decision. | ny effect ( | of the |
| Examples: a study coordinator will obtain consent instead of the subjects' physician; the not know which subjects agreed to participate; subjects will have two days to decide a the study. | | |
| e. Ongoing process. For research that involves multiple or continued interaction with subjects over the opportunities (if any) you will give subjects to ask questions or to change their minds about | | |
| There will be a single administration of the selected medication. If the participant decides that | they do n | ot wish |

to complete the VAS workbook at any time they can do so at no consequence and may return the incomplete workbook or discard it in any manner that they chose.

**8.3 Written documentation of consent.** Which of the statements below describe whether you will obtain documentation of consent? NOTE: This question does not apply to screening and recruiting procedures which have already been addressed in <u>question 4.6</u>.

Documentation of consent that is obtained electronically is not considered written consent unless it is obtained by a method that allows verification of the individual's signature. In other words, saying "yes" by email is rarely considered to be written documentation of consent

| <b>a.</b> Are you obta | ining written documentation | n of consent for: | | |
|---|---|---|---|---|
| None of y | our research procedures | → Use the table below to provide your justificati question 8.4. | on then go | to |
| X All of you | r research procedures | → Do not complete the table; go to question 8.3 | 3.b. | |
| Some of y | your research procedures | → Use the table below to identify the procedure not obtain written documentation of consent subjects. | | • |
| Adult subject<br>group¹ | | res or data/specimen collection (if any) for<br>ill be NO documentation of consent | Will<br>provide<br>with a v<br>state<br>describ<br>rese<br>(option | e them written ment ing the arch |
| <ul><li>Table footnotes</li><li>1. If your answer is the same for all adult groups or all procedures, you can collapse your answer across the groups and/or procedures.</li></ul> | | | | |
| Version 1.3 | ZIPLINE | E APPLICATION: IRB Protocol | | #2003 |

| <b>8.4 Non-English-speaking or -reading adult subjects</b> . Will you enroll adult subjects who do not speak English or who lack fluency or literacy in English? |
|---|
| <ul> <li>No</li> <li>Yes → If yes, describe the process you will use to ensure that the oral and written information provided to them during the consent process and throughout the study will be in a language readily understandable to them and (for written materials such as consent forms or questionnaires) at an appropriate reading/comprehension level.</li> </ul> |
| <b>a.</b> <u>Interpretation</u> . Describe how you will provide interpretation and when. Also, describe the qualifications of the interpreter(s) – for example, background, experience, language proficiency in English and in the other language, certification, other credentials, familiarity with the research-related vocabulary in English and the target language. |
| b. <u>Translations</u> . Describe how you will obtain translations of all study materials (not just consent forms) and how you will ensure that the translations meet the UW IRB's requirement that translated documents will be linguistically accurate, at an appropriate reading level for the participant population, and culturally sensitive for the locale in which they will be used. |
| <ul> <li>8.5 Barriers to written documentation of consent. There are many possible barriers to obtaining written documentation of consent. Consider, for example, individuals who are functionally illiterate; do not read English well; or have sensory or motor impairments that may impede the ability to read and sign a consent form.</li> <li>a. Describe your plans (if any) for obtaining written documentation of consent from potential subjects who may have difficulty with the standard documentation process (that is, reading and signing a consent form). Skip this question if you are not obtaining written documentation of consent for any part of your research.</li> </ul> |
| Examples of solutions: Translated consent forms; use of the Short Form consent process; reading the form to the person; excluding individuals who cannot read and understand the consent form. |
| I will give the participants a copy of the consent form and ask them if they would like me to read it to them or explain any portion of the form before they sign it. |
| 8.6 Deception. Will you deliberately withhold information or provide false information to any of the subjects? No Yes → If yes, describe what information and why. Example: you may wish to deceive subjects about the purpose of the study. |
| In order to have a double-blind study design, neither the subject nor the principal investigator will have knowledge of the medication that each participant will receive. |
| a. Will you debrief the subjects later? (Note: this is not required.) |
| X No Yes → If yes, describe how you will debrief the subjects. Upload any debriefing |

| _ | researd | impaired adults and other adults unable to consent. Do you plan to include such individuals in ch? |
|---|---|---|
| | | dividuals with Traumatic Brain Injury (TBI) or dementia; individuals who are unconscious, or who are intoxicated. |
| х | No | → If no, go to guestion 8.8. |
| | Yes | → If yes, answer the following questions. |
| | | <b>a.1.</b> Rationale. Provide your rationale for including this population in your research. |
| | | a.1. <u>Rationale</u> . Provide your rationale for including this population in your research. |
| | | <b>a.2.</b> Capacity for consent / decision making capacity. Describe the process you will use to determine whether a cognitively impaired individual is capable of consent decision |
| | | making with respect to your research protocol and setting. If you will have repeated interactions with the impaired subjects over a time period when cognitive capacity could increase or diminish, also describe how (if at all) you will re-assess decision-making capacity and consent during that time. |
| | | a.3. Permission (surrogate consent). If you will include adults who cannot consent for<br>themselves, describe your process for obtaining permission ("surrogate consent") from a<br>legally authorized representative (LAR). |
| | | For research conducted in Washington State, see the <b>SOP: Legally Authorized Representative</b> to learn which individuals meet the state definition of "legally authorized representative". |
| | | <b>a.4</b> . Assent. Describe whether assent will be required of all, some, or none of the subjects. If some, indicate which subjects will be required to assent and which will not (and why not). Describe any process you will use to obtain and document assent from the subjects |
| | | a.5. Dissent or resistance. Describe how you will identify the subject's objection or resistance to participation (including non-verbal) during the research, and what you will do in response. |
| consent | scripts/ | I materials. Upload to the Consent Forms and Recruitment Materials SmartForm of <i>Zipline</i> all 'talking points, consent forms, debriefing statements, Information Statements, Short Form consen permission forms, and any other consent-related materials you will use. |
| - | | must be included. However, you are strongly encouraged to wait to provide them until you know that the IR |
| | | the English versions. |
| | | forms: It may be appropriate to combine parental permission with consent, if parents are subjects as well of |

ZIPLINE APPLICATION: IRB Protocol

Version 1.3

#2003


materials, including talking points or a script, to the Consent Form and

Recruitment Materials SmartForm of *Zipline*.

(8.7)Cognitively impaired adults, and other adults unable to consent.

- providing permission for the participation of their children. Similarly, a consent form may be appropriately considered an assent form for older children.
- <u>For materials that cannot be uploaded</u>: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.

### 9 PRIVACY AND CONFIDENTIALITY

**9.1** Privacy protections. Describe the steps you will take, if any, to address possible privacy concerns of subjects and potential subjects.

Privacy refers to the sense of being in control of access that others have to ourselves. This can be an issue with respect to recruiting, consenting, sensitivity of the data being collected, and the method of data collection. Examples:

- Many subjects will feel a violation of privacy if they receive a letter asking them to participate in a study because they
  have \_\_\_\_ medical condition, when their name, contact information, and medical condition were drawn from
  medical records without their consent. Example: the IRB expects that "cold call" recruitment letters will inform the
  subject about how their information was obtained.
- Recruiting subjects immediately prior to a sensitive or invasive procedures (e.g., in an outpatient surgery waiting room) will feel like an invasion of privacy to some individuals.
- Asking subjects about sensitive topics (e.g. details about sexual behavior) may feel like an invasion of privacy to some individuals.

Patients already seeking orthodontic treatment at the University of Washington Graduate Orthodontics clinic will receive a recruitment flyer informing them of the study. If they decide they want to participate then they will receive more information.

**9.2** Identification of individuals in publications and presentations. Do you plan to use potentially identifiable information about subjects in publications and presentations, or is it possible that individual identities could be inferred from what you plan to publish or present?



- **9.3 State mandatory reporting.** Each state has reporting laws that require some types of individuals to report some kinds of abuse, and medical conditions that are under public health surveillance. These include:
  - Child abuse
  - Abuse, abandonment, neglect, or financial exploitation of a vulnerable adult
  - Sexual assault
  - Serious physical assault
  - Medical conditions subject to mandatory reporting (notification) for public health surveillance

Are you or a member of your research team likely to learn of any of the above events or circumstances while conducting your research **AND** feel obligated to report it to state authorities?

|--|

| | Yes → If yes, the UW IRB expects you to inform subjects of this possibility in the consent form or during the |
|---|---|
| | consent process, unless you provide a rationale for not doing so: |
| ider<br>afte<br>Foo<br>som<br>link | ention of identifiers and data. Check the box below to indicate your assurance that you will not destroy any natifiers (or links between identifiers and data/specimens) and data that are part of your research records until or the end of the applicable records retention requirements (e.g. Washington State; funding agency or sponsor d and Drug Administration) for your research. If you think it is important for your specific study to say nething about destruction of identifiers (or links to identifiers) in your consent form, state something like "the between your identifier and the research data will be destroyed after the records retention period required by e and/or federal law." |
| | question can be left black for conversion applications (existing paper applications that are being "converted" into a Zipline lication.) |
| recto | the "Research Data" sections of the following website for UW Records management for the Washington State research ords retention schedules that apply in general to the UW (not involving UW Medicine data): 2.//f2.washington.edu/fm/recmgt/retentionschedules/gs/general/uwgsResearch#R |
| | the "Research Data and Records" information in Section 8 of this document for the retention schedules for UW Medicine ords: <a href="http://www.uwmedicine.org/about/Documents/UWMRRS-1.5.pdf">http://www.uwmedicine.org/about/Documents/UWMRRS-1.5.pdf</a> |
| | Confirm difficates of Confidentiality. Do you have or, are you planning to obtain, a federal Certificate of Confidentiality your research data? |
| Х | No<br>Yes |
| provent<br>each<br>prot | a and specimen security protections. Identify your data classifications and the security protections you will wide, referring to the ZIPLINE GUIDANCE: Data and Security Protections for the minimum requirements for the data classification level. You cannot answer this question without reading this document. Data security tections should not conflict with records retention requirements. |
| | Which level of protections will you apply to your data and specimens? If you will use more than one level, describe which level will apply to which data and which specimens. |
| | Since this is of very low risk or harm if disclosed (level 1), no specific protections are required above and beyond standard University expectations. |
| | Use this space to provide additional information, details, or to describe protections that do not fit into one of the levels. |
| | No identifiers will be made on the workbook materials that each participant will return. Contact information for reminder notifications will be stored in a locked computer file that is separate than the data file. |
| | Upon completion, the participant can elect to enter a raffle by writing their contact information on a ticket and place it into a locked box that will be stored securely behind the front office of the clinic. No information pertaining to the study will be discerned from the raffle ticket except for the fact that that individual has |

#2003

completed a workbook for the study.

### **10 RISK / BENEFIT ASSESSMENT**

- **10.1**) Anticipated risks. Describe the <u>reasonably foreseeable</u> risks of harm, discomforts, and hazards to the subjects and others of the research procedures. For each harm, discomfort, or hazard:
  - Describe the magnitude, probability, duration, and/or reversibility of the harm, discomfort, or hazard, AND
  - Describe how you will manage or reduce the risks. Do not describe data security protections here, these are already described in Question 9.6.
  - Consider physical, psychological, social, legal, and economic risks, including risks to financial standing, employability, insurability, educational advancement or reputation.
  - Examples of "others": embryo, fetus, or nursing child; family members; a specific group.
  - Do not include the risks of non-research procedures that are already being performed.
  - If the study design specifies that subjects will be assigned to a specific condition or intervention, then the condition or intervention is a research procedure even if it is a standard of care.
  - Examples of mitigation strategies: inclusion/exclusion criteria; applying appropriate data security measures to prevent unauthorized access to individually identifiable data; coding data; taking blood samples to monitor something that indicates drug toxicity.
  - As with all questions on this application, you may refer to uploaded documents.

Reactions or adverse effects of the medications involved are known and may occur in the subjects. All subjects will be assessed to ensure they are not contraindicated for these medications. The consent form will outline possible adverse effects and will be made known to the subjects prior to initiation of the study.

The following are adverse reacts associated with the involved medications and typically occur when the medications used at high doses or chronically in <10% of the population:

- Anemia
- Kidney failure
- Liver failure
- Edema
- Dizziness
- Blurred vision
- Headache
- Rash
- Heartburn
- Nausea
- Cardiovascular thrombotic events
- Ulcers
- Bronchospasms

Reproductive risks. Are there any risks of the study procedures to men and women (who are subjects, or partner of subjects) related to pregnancy, fertility, lactation or effects on a fetus or neonate?

Examples: direct teratogenic effects; possible germline effects; effects on fertility; effects on a woman's ability to continue a pregnancy; effects on future pregnancies.

x

No  $\rightarrow$  If no go to guestion 10.3

Vac

→ If yes, answer the following questions:

a. Risks. Describe the magnitude, probability, duration and/or reversibility of the risks.

Ibuprofen used in late pregnancy should be avoided due possible causation of premature closure of the ductus arteriosus.


| | <b>b. Steps to minimize risk</b> . Describe the specific steps you will take to minimize the magnitude, probability, or duration of these risks. |
|---|---|
| | Examples: inform the subjects about the risks and how to minimize them; require a pregnancy test before and during the study; require subjects to use contraception; advise subjects about banking of sperm and ova. |
| | If you will require the use of contraception: describe the allowable methods and the time period when contraception must be used. |
| | Female participants that are pregnant will be excluded from the study. |
| | c. Pregnancy. Describe what you will do if a subject (or a subject's partner) becomes pregnant |
| | For example; will you require the subject to immediately notify you, so that you can discontinue or modify the study procedures, discuss the risks, and/or provide referrals or counseling? |
| | The study requires only a single administration of a medication at the initiation of the study so there will be no risk if the subject becomes pregnant afterwards. |
| 10.3 Unforeseea | ble risks. Are there any research procedures that may have risks that are currently unforeseeable? |
| No | ng a drug that hasn't been used before in this subject population. If yes, identify the procedures. |
| <u> </u> | In the highly unlikely event that a patient has an unknown hypersensitivity to one of the medications, associated risks of hypersensitivities may occur. |
| anesthesia X No | tients are under general or regional anesthesia, or during the 3 hours preceding general or regional (supplied for non-research reasons)? → If yes, check all the boxes that apply. |
| | Administration of any drug for research purposes |
| | Inserting an intra-venous (central or peripheral) or intra-arterial line for research purposes |
| | Obtaining samples of blood, urine, bone marrow or cerebrospinal fluid for research purposes |
| | Obtaining a research sample from tissue or organs that would not otherwise be removed during surgery |
| | Administration of a radio-isotope for research purposes** |
| | Implantation of an experimental device |
| | Other manipulations or procedures performed solely for research purposes (e.g., experimental liver dialysis, experimental brain stimulation) |

| If you checked any of the boxes: |
|---|
| You must provide the name and institutional affiliation of a physician anesthesiologist who is a |
| member of your research team or who will serve as a safety consultant about the interactions |
| between your research procedures and the general or regional anesthesia of the subject- |
| patients. If your procedures will be performed at a UW Medicine facility or affiliate, the |
| anesthesiologist must be a UW faculty member. |

\*\* If you checked the box about radio-isotopes: you are responsible for informing in advance all appropriate clinical personnel (e.g., nurses, technicians, anesthesiologists, surgeons) about the administration and use of the radio-isotope, to ensure that any personal safety issues (e.g., pregnancy) can be appropriately addressed. This is a condition of IRB approval.

**10.5 Data and Safety Monitoring**. A Data and Safety Monitoring Plan (DSMP) is required for clinical trials (as defined by NIH). If required for your research, upload your DSMP to the **Supporting Documents** SmartForm in **Zipline**. If it is embedded in another document you are uploading (for example, a Study Protocol, use the text box below to name the document that has the DSMP.

N/A

**10.6 Un-blinding.** If this is a double-blinded or single-blinded study in which the participant and/or you do not know the group to which the participant is assigned: describe the circumstances under which un-blinding would be necessary, and to whom the un-blinded information would be provided.

If a patient has an allergic response to their medication, they will be made aware of which medication they were administered.

**10.7 Withdrawal of participants.** If applicable, describe the anticipated circumstances under which participants will be withdrawn from the research without their consent. Also, describe any procedures for orderly withdrawal of a participant, regardless of the reason, including whether it will involve partial withdrawal from procedures and any intervention but continued data collection or long-term follow-up.

N/A

Anticipated direct benefits to participants. If there are any direct research-related benefits that some or all individual participants are likely to experience from taking part in the research, describe them below:

Do not include benefits to society or others, and do not include subject payment (if any). Examples: medical benefits such as laboratory tests (if subjects receive the results); psychological resources made available to participants; training or education that is provided.

Analgesia for pain induced by orthodontic tooth movement.

- 10.9 Individual subjects findings.
  - **a**. Is it likely that your research will unintentionally discover a previously unknown condition such as a disease, suicidal intentions, or genetic predisposition?

X No

→ If yes, explain whether and how you would share the information with the subject.

| genetic test results, laboratory tests, etc.? X No Yes If yes, complete and upload the SUPPLEMENT: Participant Results Sharing to the Supporting Documents SmartForm of Zipline |
|---|
| 10.10 Commercial products or patents. If a commercial product or patent could result from this study, describe whether subjects might receive any remuneration/compensation and, if yes, how the amount will be determined: |
| N/A |
| 11 ECONOMIC BURDEN TO PARTICIPANTS |
| <b>11.1 Financial responsibility for research-related injuries.</b> Answer this question only if the lead researcher is <u>not</u> a UW student, staff member, or faculty member whose primary paid appointment is at the UW. |
| Describe who will be financially responsible for research-related injuries experienced by subjects, and any limitations. Describe the process (if any) by which participants may obtain treatment/compensation. |
| N/A |
| 11.2 Costs to subjects. Describe any research-related costs for which subjects may be responsible (e.g., CT scan required for research eligibility screening; co-pays; cost of a device; travel and parking expenses that will not be reimbursed). |
| None. |
| 11.3 Reimbursement for costs. Describe any costs to subjects that will be reimbursed (such as travel expenses). |
| None. |
| 12 RESOURCES |
| Faculty Advisor. (For researchers who are students, fellows, or post-docs.) Provide the following information about your faculty advisor. • Advisor's name |
| <ul> <li>Your relationship with your advisor (for example: graduate advisor; course instructor)</li> <li>Your plans for communication/consultation with your advisor about progress, problems, and changes.</li> </ul> |
| Dr. Anne-Marie Bollen<br>Research Advisor<br>Dr. Bollen is regularly available in the clinic in which the study will take place. |
| ZIPLINE APPLICATION: IRB Protocol #2003 Version 1.3 |


| <b>12.2 Study team communication</b> . Describe how you will ensure that each study team member is adequately trained and informed about the research procedures and requirements (including any changes) as well as their research related duties and functions. | |
|---|---|
| There is no study team. | |
| 13 OTHER APPROVALS, PERMIS | SSIONS, and REGULATORY ISSUES |
| <b>13.1 Other regulatory approvals</b> . Identification checking applicable boxes | fy any other regulatory approvals that are required for this research, by |
| Do not attach the approvals unless requ | ested by the IRB. |
| Approval | Research for which this is required |
| Radiation Safety | Procedures involving the use of radioactive materials or an ionizing radiation producing machine radiation, if they are conducted for research rather than clinical purposes. Approvals need to be attached to the Supporting Documents page in <i>Zipline</i> . |
| Institutional Biosafety | Procedures involving the transfer/administration of recombinant DNA, DNA/RNA derived from recombinant DNA, or synthetic DNA. |
| RDRC | Procedures involving a radioactive drug or biological product that is not approved by the FDA for the research purpose and that is being used without an IND, for basic science research (not to determine safety and effectiveness, or for immediate therapeutic or diagnostic purposes). |
| ESCRO | Procedures involving the use of some types of human embryonic stem cells. |
| | y any other approvals or permissions that will be obtained. For example: ation, funding agency, employee union, UW Medicine clinical unit. |
| Do not attach the approvals and permissions unless requested by the IRB. | |
| N/A | |
| Financial Conflict of Interest. Does research, as defined by UW policy C | any member of the team have a Financial Conflict of Interest (FCOI) in this <u>GIM 10</u> ? |
| Yes → If yes, upload the Conflict Management Plan for every team member who has a FCOI with respect to this research, to the <b>Supporting Documents</b> page of <b>Zipline</b> . If it is not yet available, use the text box to describe whether the Significant Financial Interest has been disclosed already to the UW Office of Research. | |
| | ZIPLINE APPLICATION: IRB Protocol #2003 |


Version 1.3